CLINICAL TRIAL: NCT00139178
Title: Switching From Zidovudine to an NNRTI or Lopinavir/Ritonavir in Patients Treated With Zidovudine/ Lamivudine/Abacavir. Influence on Metabolic Abnormalities
Brief Title: Switching From Zidovudine to an NNRTI or Lopinavir/Ritonavir in Patients Treated With Zidovudine/ Lamivudine/Abacavir.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danish HIV Research Group (Other)
Collaborators: Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Aarhus University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26122450
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-08

CONDITIONS: HIV Associated Lipodystrophy Syndrome.; HIV; Hypercholesterolemia; Lipoatrophy
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Hypercholesterolemia; Lipodystrophy

INTERVENTIONS:
Drug: Different HAART regimens

SUMMARY:
Highly active antiretroviral therapy (HAART) has improved the long time survival of HIV infected individuals. However an increasing number of HIV-patients have developed metabolic and morphological alterations including peripheral lipoatrophy.

The main hypothesis of the study is that switching from thymidine-analogue based HAART will reverse lipoatrophy.

We plan to perform an observational study recruiting up to 100 HIV-infected patients receiving Trizivir (zidovudine/lamivudine/abacavir).

The patients will be offered an NRTI or lopinavir/ritonavir instead of zidovudine or they can choose to continue with Trizivir.

The main endpoint is changes in peripheral fat mass as determined by DEXA-scanning.

ELIGIBILITY:
Inclusion Criteria:

* Currently treated with lamivudine, zidovudine and abacavir
* Viral load < 200 copies/ml
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Women being pregnant or breast-feeding.
* Fertile women using no safe contraception.
* Patients with active intravenous drug use.
* Abuse of alcohol, which in the opinion of the treating physician will reduce the patient´s ability to follow a therapeutic regimen and evaluations of the protocol.
* Creatinine > 200 mmol/l.
* ALT or AST > 5 times upper normal value (200U/l).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-03; Study Completion 2007-04

PRIMARY OUTCOMES:
Changes in peripheral fat mass, determined by DEXA-Changes Change from baseline in fasting lipids and subsets hereof. Development of impaired glucose tolerance and insulin resistance.

SECONDARY OUTCOMES:
Changes in body composition from baseline, determined by patient and physician in a standardized questionnaire and by standardized clinical examination.
Proportion of patients with HIV-RNA < 20 copies after 24, 48, 72 and 96 weeks.
Change in CD4 cell count from baseline after 24, 48, 72 and 96 weeks.
Incidence of adverse events.
Incidence of clinical disease progression.
Proportion of patients who have virological, immunological or clinical failure or treatment-limiting adverse events at week 24,48 and 96.
Change in plasma lactate from baseline.
Time to discontinuation of the allocated therapy and reasons for this.
Incidence of genotypical and virological resistance. Development of osteopenia, judged by DEXA-scan. Compliance - proportion of patients who report to take 90%, respectively 95% of their medications at week 4, 48 and 96.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gerstoft, M.D., DMSc, Principal Investigator — Rigshospitalet, Denmark; Ann-Brit E Hansen, M.D., Principal Investigator — Odense University Hospital; Court Pedersen, Professor, Principal Investigator — Odense University Hospital; Lars Mathiesen, M.D. DMSc, Principal Investigator — Hvidovre University Hospital; Alex Laursen, D.M., DMSc, Principal Investigator — Aarhus University Hospital; Niels Obel, Study Chair — Odense University Hospital
Locations (4):
- Denmark (4):
  - Department of Infectious Diseases, Aarhus University Hospital, Aarhus
  - Department of Infectious Diseases, Rigshospitalet, Copenhagen
  - Department of Infectious Diseases, Hvidovre University Hospital, Hvidovre
  - Department of Infectious diseases, Odense University Hospital, Odense